CLINICAL TRIAL: NCT06309095
Title: Investigation of the Effect of Low Torque and Speed on Post-Operative Pain After Root Canal Treatment: A Randomized Clinical Study
Brief Title: Investigation of the Effect of Low Torque and Speed on Post-Operative Pain After Root Canal Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Ahmet Demirhan Uygun, Associate Professor, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AFSU_AhmetDemirhanUygun_001
Record Dates: First submitted 2024-02-21; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Dental Pulp Necrosis
Keywords: Devital tooth
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1 N (Newton) torque, 250 rpm(rotary per minute) speed (Experimental): The values specified in the endomotor will be used during root canal treatment. 1 N torque, 250 rpm speed
  Interventions: Device: use of VDW Silver Endodontic motor
- 1 N torque, 350 rpm speed (Experimental): The values specified in the endomotor will be used during root canal treatment. 1 N torque, 350 rpm speed
  Interventions: Device: use of VDW Silver Endodontic motor
- 2 N torque, 250 rpm speed (Experimental): The values specified in the endomotor will be used during root canal treatment. 2 N torque, 250 rpm speed
  Interventions: Device: use of VDW Silver Endodontic motor
- 2 N torque, 350 rpm speed (Experimental): The values specified in the endomotor will be used during root canal treatment. 2 N torque, 350 rpm speed
  Interventions: Device: use of VDW Silver Endodontic motor

INTERVENTIONS:
Device: use of VDW Silver Endodontic motor — All patients will be subjected to local anesthesia with articaine hydrochloride (Maxicaine, Istanbul) containing 1:100,000 adrenaline. After the entrance cavities of the teeth are opened, a rubber dam will be applied to the relevant teeth for isolation from the oral environment. After the entrance cavity is opened, the working length of the canals will be determined with the help of a No. 10 K-file (Dentsply Maillefer, Ballaigues, Switzerland) canal file and an electronic apex finder (Woodpex III, Woodpecker Medical Instrument Co, Guilin, China). In both groups, it was planned to use the NiTi rotary instrument system using V Taper Gold (Fanta Dental Material, Shanghai, China) files with the help of VDW.Silver endomotor (VDW, München, Germany). The endodontic motor will be used to adjust different speed and torque values during root canal treatment. Post-operative pain caused by different speed and torque values will be compared.

SUMMARY:
Root canal preparation is one of the most important stages in root canal treatment. Nowadays, the use of Nickel-Titanium(Ni-Ti) rotary instrument systems for root canal expansion is becoming very popular. The force required to rotate the Ni-Ti file is defined as the torque force and is considered a parameter for the stress produced within the canal. Ni-Ti rotary instruments can be used with a wide speed scale between 150 rpm (rotary per minute) and 40,000 rpm in conventional endodontic engines.

Low torque and speed values mean low pressure applied by the instruments in the root canal. With low forces and vibrations, motor noise is generally negligible, and the instruments can easily shape most root canals in a reasonable amount of time and with minimal mechanical stress (in medium-easy canals). The use of lower torque values has been shown to reduce cyclic fatigue of Ni-Ti rotary tools. With reduced cyclic fatigue, the risk of instrument breakage in complex root canal morphologies is minimized and complications that may occur during root canal treatment are reduced. However, with low torque and speed values, cutting efficiency decreases and the process time increases as the instrument advances in the canal and during possible treatment. Decreasing cutting efficiency may also result in the operator applying force to move through the canal. With the applied force, the friction resistance within the canal increases and the heat produced increases. For this reason, it is thought that the risk of post-operative pain may increase during or after the procedure.

The aim of this study is to investigate the incidence of post-operative pain and procedure time using the visual analog scale (VAS) among groups where low torque and speed values were applied during the use of the Ni-Ti rotary instrument system.

DETAILED DESCRIPTION:
Patients with an indication for root canal treatment of the mandibular first molar tooth, who applied to Faculty of Health Sciences, Department of Endodontics, were selected. Patients aged between 18 and 65, who volunteered for the study and had no systemic disease and no preoperative pain, were included.

Patients meeting the inclusion criteria will be randomly divided into four groups (n=20) using a website (www.randomizer.org). The patient number and the randomized group from which the patient was selected will be recorded. All patients will be subjected to local anesthesia with articaine hydrochloride (Maxicaine, Istanbul) containing 1:100,000 adrenaline. After the entrance cavities of the teeth are opened with an aerator under water cooling, a rubber dam will be applied to the relevant teeth for isolation from the oral environment. After the entrance cavity is opened, the working length of the canals will be determined with the help of a No. 10 K-file (Dentsply Maillefer, Ballaigues, Switzerland) canal file and an electronic apex finder (Woodpex III, Woodpecker Medical Instrument Co, Guilin, China). In both groups, it was planned to use the NiTi rotary instrument system using V Taper Gold (Fanta Dental Material, Shanghai, China) files with the help of VDW.Silver endomotor (VDW, München, Germany). The patient groups were determined as the first group was 2N torque value and 350 rpm speed, the second group was 2N torque and 250 rpm speed, the third group was 1N torque and 350 rpm speed, and the fourth group was 1N torque and 250 rpm speed. The torque values to be applied are lower than the values recommended by the manufacturer and there is no harm in applying them in the literature. For irrigation of root canals, 2ml of 2.5% sodium hypochlorite will be used at each instrument change. For final irrigation, 17% EDTA( ethylenediaminetetraacetic acid) solution will be used. Root canals will be dried using sterile paper points. The root canals will be filled using gutta percha and a resin-containing root canal sealer (Dentsply Maillefer, Ballaigues, Switzerland) and the treatment will be completed by making the upper restoration. After the treatment, patients were given a VAS scale (Visual Analog Scale) and were instructed how to fill in their pain levels verbally and visually, 6, 12, 48, 72 hours and 1 week later. With the VAS scale, patients will be asked to note whether they use the prescribed Ibuprofen analgesic and the frequency of use. When patients come to their follow-up appointment, the forms will be taken from the patients and their post-treatment pain values will be compared. The collected data will be analyzed statistically with one-way ANOVA and post hoc Tukey tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients without a history of intolerance to nonsteroidal anti-inflammatory drugs
* Patients who have no physical or psychological disabilities and are competent in understanding and applying treatment protocols
* Mandibular first molars without preoperative pain,
* The relevant tooth is devital (non-living)
* Teeth that have not had root canal treatment before,
* Teeth that have not been traumatized and have no serious dental malposition,
* Teeth that do not have complex root canal morphology,
* Patients whose root curvature is not >25°,
* Patients without sinus tract, periapical abscess and cellulitis,

Exclusion Criteria:

* Pregnancy and patients who may be pregnant
* Patients who have used cortisone in the last 6 months and analgesic-anti-inflammatory-antibiotic use in the last week
* The patient is allergic to one or more of the agents to be used during the procedure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale | through study completion, an average of 1 month
  The patient was asked to mark the severity of his or her pain with active motion on a horizontal line 100 mm in lenght. The intensity of the pain was calculated by measuring the area in which the individual marked between 0 (no pain) and 10 (the most severe pain I felt my life)

SECONDARY OUTCOMES:
Preparation time | through study completion, an average of 1 month
  While shaping the root canals at the specified values, the working time (second) will be measured with the help of a stopwatch.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet D Uygun, Assoc. Prof., Study Chair — Afyonkarahisar Health Science University/ Dentistry Faculty
Locations (1):
- Afyonkarahisar Health Science University, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No